CLINICAL TRIAL: NCT06871891
Title: Effect of Perioperative Sleep Quality on Chronic Post-Surgical Pain: a Prospective Cohort Study
Brief Title: Effect of Perioperative Sleep Quality on Chronic Post-Surgical Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); National Cancer Center/National Cancer Clinical Medical Research Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College (Unknown)
Responsible Party: Principal Investigator, Lu Che, Attending Anesthesiologist, Peking Union Medical College Hospital
Other Study IDs: K7648
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Chronic Post-Surgical Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SLEEP-CPSP Cohort

SUMMARY:
The goal of this prospective observational cohort study is to assess the impact of perioperative sleep quality on the development of chronic post-surgical pain (CPSP) in adult patients (aged 18-80 years, ASA I-III) undergoing elective video-assisted thoracic surgery (VATS), modified radical mastectomy (MRM), or coronary artery bypass grafting (CABG). The main questions it aims to answer are:

Does poor perioperative sleep quality increase the risk of CPSP at 3 months post-surgery? How do subjective and objective sleep parameters (e.g., total sleep duration, deep sleep time) correlate with CPSP and recovery outcomes? Researchers will compare patients with varying perioperative sleep quality levels (assessed via the Richards-Campbell Sleep Questionnaire [RCSQ] and wearable device data) to evaluate differences in CPSP incidence, pain and quality of life.

Participants will:

Wear a Huawei wearable device to collect objective sleep data (e.g., sleep duration, deep sleep time) during hospitalization.

Complete questionnaires preoperatively and postoperatively, including RCSQ, Pittsburgh Sleep Quality Index (PSQI), Hospital Anxiety and Depression Scale (HADS), and Brief Pain Inventory (BPI).

Undergo follow-up assessments at 1, 3, and 6 months post-surgery to evaluate pain scores , CPSP status, and quality of life (SF-36).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years.
2. Scheduled for elective video-assisted thoracic surgery (VATS).
3. Scheduled for elective modified radical mastectomy (MRM).
4. Scheduled for elective coronary artery bypass grafting (CABG).
5. American Society of Anesthesiologists (ASA) physical status classification I-III.
6. Willing to sign the informed consent form, participate in the study, and complete all follow-up assessments.

Exclusion Criteria:

1. History of surgery within the past 3 months.
2. Chronic use of opioids or sedatives (defined as use for 3 months or longer).
3. Expected completion time of surgery after 16:00 on the day of operation.
4. Planned transfer to the intensive care unit (ICU) postoperatively.
5. Anticipated hospital stay <24 hours.
6. Contraindications to wearable device use (e.g., infection at the wrist site, allergy to the wristband material).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from Peking Union Medical College Hospital, Fuwai Hospital, and Cancer Hospital to reflect diverse clinical practices.
Sampling Method: Non-Probability Sample
Enrollment: 1138 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
chronic post-surgical pain (CPSP): Brief Pain Inventory (BPI) | at 3 months after surgery
  The Brief Pain Inventory (BPI) is a widely used pain assessment tool for evaluating pain intensity and impact, suitable for chronic pain patients. It measures current, least, worst and average pain in the past 24 hours on a 0 - 10 scale (0=no pain, 10=extreme pain), and assesses pain's effect on 7 daily life aspects, scored 0 - 10 (0=no interference, 10=total interference). If a participant's BPI evaluation shows a pain condition and also meets these five criteria: (1) Pain arises or intensifies following surgery; (2) Pain persists for at least three months and impacts quality of life; (3)Pain occurs after a pain-free interval or evolves from ongoing acute postoperative pain; (4) Pain is localized to the surgical site or radiates to areas corresponding to the relevant nerve distribution; and (5) Other potential causes of pain are excluded.
Subjective sleep assessment: Richards - Campbell Sleep Questionnaire (RCSQ) | 1 day before surgery and 1st, 2nd, and 3rd days after surgery.
  The Richards-Campbell Sleep Questionnaire (RCSQ) is a prominent tool in sleep research and clinical practice for gauging sleep quality. It comprehensively evaluates sleep aspects from respondents' subjective views. Comprising multiple items, it covers sleep onset latency (time to fall asleep), sleep depth, sleep duration, and wake-up frequency at night. It may also involve related factors like sleep environment quality and sleep's impact on daily life. With specific questions and response options, individuals rate sleep experiences numerically or descriptively. Data from the RCSQ aids in diagnosing sleep disorders, evaluating treatment efficacy, and conducting sleep-related epidemiological studies. It is mainly intended for the assessment of short-term sleep conditions during hospitalization.

SECONDARY OUTCOMES:
Pain assessment: Numerical rating scale (NRS) | 1st, 2nd, 3rd days after surgery and at 1 months after surgery
  The Numerical Rating Scale (NRS) for pain is a commonly used tool in healthcare to gauge patients' pain intensity. It's a subjective measure where patients rate pain on a 0 - 10 scale. 0 means no pain; 10 is the worst imaginable pain. Scores 3 and below suggest mild pain with little impact, 4 - 6 moderate pain affecting daily life somewhat, and 7 and above severe pain needing prompt attention. It's practical for its simplicity. Medical staff can administer it quickly during consultations. Patients can easily understand and use it to convey pain feelings. This helps professionals evaluate pain severity, plan treatments, and monitor pain relief. Overall, the NRS is vital in pain assessment and management, enhancing medical care quality and patient comfort.
chronic post-surgical pain (CPSP) : Brief Pain Inventory (BPI) | at 6 months after surgery
  The Brief Pain Inventory (BPI) is a widely used pain assessment tool for evaluating pain intensity and impact, suitable for chronic pain patients. It measures current, least, worst and average pain in the past 24 hours on a 0 - 10 scale (0=no pain, 10=extreme pain), and assesses pain's effect on 7 daily life aspects, scored 0 - 10 (0=no interference, 10=total interference). If a participant's BPI evaluation shows a pain condition and also meets these five criteria: (1) Pain arises or intensifies following surgery; (2) Pain persists for at least three months and impacts quality of life; (3)Pain occurs after a pain-free interval or evolves from ongoing acute postoperative pain; (4) Pain is localized to the surgical site or radiates to areas corresponding to the relevant nerve distribution; and (5) Other potential causes of pain are excluded.
Quality of life assessment: Short Form-36 Health Survey Questionnaire (SF-36) | 1, 3, 6 months after surgery
  Short Form-36 Health Survey Questionnaire (SF-36) The SF-36 is a widely recognized and commonly used instrument for assessing quality of life. It consists of 36 questions covering eight domains, such as physical functioning, role limitations due to physical problems, social functioning, and mental health.The scale provides a comprehensive view of an individual's quality of life, generating scores that help healthcare providers understand patients' well-being and make more informed decisions in diagnosis, treatment, and care, with good reliability and validity demonstrated in various studies.
Quality of recovery assessment: Quality of Recovery-15 (QoR-15) assessment scale | 1st and 3rd days after surgery
  The Quality of Recovery-15 (QoR-15) assessment scale is a professional tool for evaluating the recovery quality of patients post-surgery or after certain medical interventions. It is composed of 15 items, with each item scored from 0 to 10 points, and the total score ranges from 0 to 150 points. The higher the score, the better the quality of recovery. These 15 items cover five dimensions: physical comfort, emotional state, physical independence, psychological support, and pain. The QoR-15 scale is recognized for its high reliability and validity. It is easy to administer and score, which is of great significance in assessing patients' recovery status and guiding medical staff to formulate appropriate treatment and care plans.
Subjective sleep assessment: Pittsburgh Sleep Quality Index (PSQI) | 1, 3, and 6 months after surgery.
  The Pittsburgh Sleep Quality Index (PSQI), developed by Dr. Daniel J. Buysse and his colleagues at the University of Pittsburgh in 1989, contains 19 self-rated and 5 observer-rated questions grouped into 7 components including subjective sleep quality and sleep latency etc., with each component scored 0 - 3 and total score 0 - 21, where 5 or less means good sleep quality and 5 or more indicates poor sleep quality, and it's widely used in sleep medicine, psychology and clinical research to evaluate sleep problems, monitor treatment effects and conduct epidemiological investigations, being a reliable and valid tool for assessing sleep quality and crucial for understanding and managing sleep-related issues.

OTHER OUTCOMES:
Objective sleep assessment: Total sleep duration, wake - up time during sleep, and deep sleep time. | Preoperative day 1 (the night before surgery), the night of surgery (postoperative day 0), and postoperative days 1, 2, and 3
  We will use Huawei smart wearable devices to assess the objective sleep conditions of patients. The definition of total sleep duration is as follows: Before the sleep on the first night before their surgery, a wearable sleep monitoring device was placed on the non-dominant wrist of each participant. The patients wore this sleep monitoring device throughout their hospitalization. The sleep monitoring period is from 20:00 to 20:00 the next day. The indicator of Wake-up time during sleep refers to the total time a person is awake after initially falling asleep. The deep sleep duration: According to Huawei's scientific sleep (TruSleep™) technology, the sleep status of patients is determined by analyzing data such as the patients' heart rate and body movements, and it is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
ndividual participant data (including demographic, clinical, and sleep monitoring data) will not be made publicly available to protect participant privacy and comply with ethical regulations.